CLINICAL TRIAL: NCT01422317
Title: Effects of a High-dose Concentrate of n-3 Fatty Acids or Corn Oil Introduced Early After an Acute Myocardial Infarction on Serum Triacylglycerol and High-density Lipoprotein (HDL)- Cholesterol
Brief Title: Effects of High-dose n-3 Fatty Acids on Clinical Outcome and Serum Lipids - Omacor Following Acute Myocardial Infarction
Acronym: OFAMI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Helse Stavanger HF (Other Government)
Collaborators: University of Bergen (Other); University of Oslo (Other); Pharmacia and Upjohn (Industry); Pronova BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OFAMI1995
Record Dates: First submitted 2011-08-18; First posted 2011-08-23 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Coronary Disease; Myocardial Infarction
Keywords: n-3 fatty acids; randomized double-blind study; coronary events; serum lipids; antithrombotic effects of omega-3 fatty acids; anti-inflammatory effects of omega-3 fatty acids; prognostic biomarkers in myocardial infarction (MI)-patients
MeSH Terms: conditions — Coronary Disease; Myocardial Infarction | interventions — alpha-Tocopherol; Corn Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- n-3 fatty acids (Experimental): Two gelatine capsules of Omacor-R (Pronova AS, Oslo) twice a day, each capsule containing eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA) as ethylesters, in the average ratio of EPA to DHA of 1:2. Alpha-Tocopherol (4 mg) was added to each capsule.
  Interventions: Drug: EPA / DHA / Alpha-Tocopherol
- Corn Oil (Active Comparator): Two gelatine capsules twice a day, each containing 1 gram of corn oil. Alpha-Tocopherol (4 mg) was added to each capsule.
  Interventions: Drug: EPA / DHA / Alpha-Tocopherol; Drug: Corn Oil / Alpha-Tocopherol (4 mg)

INTERVENTIONS:
Drug: EPA / DHA / Alpha-Tocopherol — Two gelatine capsules of Omacor-R (Pronova AS, Oslo) twice a day, each containing 850-882 mg eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA) as ethylesters in the average ratio of EPA to DHA of 1:2. Alpha-Tocopherol (4 mg) was added to each capsule.
  Other Names: Omacor-R
Drug: Corn Oil / Alpha-Tocopherol (4 mg) — Two gelatine capsules twice a day. Each capsule contains 1g Corn Oil and 4 mg Alpha-Tocopherol
  Other Names: Corn oil
  Arms: Corn Oil

SUMMARY:
The object of this study was to evaluate the effect of a high-dose ethylester concentrate of of n-3 fatty acids administered early after an acute myocardial infarction on subsequent cardiac events and serum lipids.The second purpose of this study was to assess the impact of high-dose n-3 fatty acids on several markers of coagulation, inflammation, endothelial dysfunction and lipid peroxidation. Re-investigation was intended after a prolonged wash-out-period.

DETAILED DESCRIPTION:
Results of epidemiologic studies and clinical trials indicate that moderate doses of n-3 unsaturated fatty acids reduce the risk of cardiovascular disease(CVD) and may improve prognosis. N-3 fatty acids have several beneficial cardiovascular properties (1-3), including antiatherothrombotic, antiarrhythmic, and antihypertensive effects, and are especially noted for their triacylglycerol-reducing ability (3-7). These effects may translate into an improved clinical outcome in patients with coronary artery disease (CAD) (8).

The pronounced effect obtained of moderate doses of n-3 fatty acids supplementation may suggest an even stronger effect of pharmacologic doses.

The object of this study was therefore to assess the effect of a high-dose ethylester concentrate of n-3 fatty acids as compared to corn oil administered early (4-8 days) after an acute myocardial infarction (MI), on fatal and non-fatal subsequent cardiac events (cardiac death, resuscitation, recurrent myocardial infarction (MI) or angina pectoris), during 2 ys follow-up (median 18 months). We hypothesized that a high-dose of n-3 fatty acids would improve serum lipids in this population, and beneficially influence several markers of coagulation, endothelial dysfunction and inflammation.

Three hundred patients with an acute myocardial infarction (MI) were recruited at one hospital center (Central Hospital in Rogaland, Stavanger, Norway) from September 1995 until December 1996. All patients were included between the fourth and the eighth day after an acute myocardial infarction (MI). All patients were randomly assigned to receive 2 gelatin capsules of Omacor-R (Pronova AS, Oslo) or corn oil twice a day. Each capsule contained either 850-882 mg eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA) as ethylesters in the average ratio of eicosapentaenoic acid (EPA) to docosahexaenoic acid (DHA) of 1:2 or the same amount of corn oil. α-Tocopherol (4 mg) was added to all capsules. The capsules were administered in a double-blind manner over 12-24 months. A detailed patient history was recorded and a clinical examination was performed. The electrocardiogram was scrutinized for infarct location. The recent injury was classified as an anterior or inferior Q-wave infarction or any non-Q-wave infarction. Treatment was initiated immediately after inclusion and collection of baseline blood samples. The study was approved by the Regional Ethics Committee for Western Norway.

Clinical follow-up, including blood tests and electrocardiogram recordings, was repeated at 6 wk, 6 mo, 1 y, 18 mo, and, for some patients, 2 ys after the start of treatment. A deviation of 2 wk at the first follow-up and ≤1 mo at later follow-ups was allowed. All cardiac events and ongoing medication were recorded. Cardiac events were defined as cardiac death, resuscitation, recurrent myocardial infarction (MI), and unstable angina. Revascularization and death from other causes were also recorded. The study was closed at the end of 1997. The median follow-up time (ignoring events except deaths) was 1.5 y.

Analyses of serum triacylglycerols, total cholesterol and high-density lipoprotein (HDL)-cholesterol were performed at inclusion, 6 weeks, 6 and 12 months. In addition, analyses of markers of inflammation [high-sensitivity-C-reactive protein (CRP), CD-40 Ligand (CD40L)], coagulation [D-Dimer, fibrinogen, tissue factor, activated factor XII (FXIIa)], endothelial dysfunction [adhesion molecules such as E-selectin and Intra-Cellular Adhesion Molecule-1 (ICAM-1), homocysteine)], and Thiobarbituric Acid Reactive Substances (TBARS) as a marker of the oxidative burden of n-3 fatty acids, have been performed at different time points during follow-up, to evaluate the influence of n-3 fatty acids on these markers, and to assess their prognostic ability following a myocardial infarction (MI). Moreover, holo-transcobalamin (holoTC), methylmalonic acid (MMA), n-Terminal pro-Brain Natriuretic Peptide (NT-proBNP), matrix metalloproteinases-9 (MMP-9), Pregnancy-associated plasma protein A (PAPP-A), myeloperoxidase (MPO), and CD40 Ligand (CD40L) were measured also in order to evaluate their prognostic ability following a myocardial infarction (MI).

After closure of the main study, the purpose was to evaluate the prognosis of the study subjects after a prolonged wash-out period.

Publications from the study:

1. Nilsen DWT, Albrektsen G, Landmark K, Moen S, Aarsland T, Woie L. Effects of a high-dose concentrate of n-3 fatty acids or corn oil introduced early after an acute myocardial infarction on serum triacylglycerol and HDL cholesterol. Am J Clin Nutr 2001;74:50-6.
2. Grundt H, Nilsen DW, Mansoor MA, Hetland Ø, Nordøy A. Reduction in homocysteine by n-3 polyunsaturated fatty acids after 1 year in a randomised double-blind study following an acute myocardial infarction: no effect on endothelial adhesion properties. Pathophysiol Haemost Thromb. 2003 Mar-Apr;33(2):88-95.
3. Grundt H, Nilsen DW, Mansoor MA, Nordøy A. Increased lipid peroxidation during long-term intervention with high doses of n-3 fatty acids (PUFAs) following an acute myocardial infarction. Eur J Clin Nutr. 2003 Jun;57(6):793-800.
4. Grundt H, Hetland Ø, Nilsen DW. Changes in tissue factor and activated factor XII following an acute myocardial infarction were uninfluenced by high doses of n-3 polyunsaturated fatty acids. Thromb Haemost. 2003 Apr;89(4):752-9.
5. Grundt H, Nilsen DW, Hetland Ø, Mansoor MA. Clinical outcome and atherothrombogenic risk profile after prolonged wash-out following long-term treatment with high doses of n-3 PUFAs in patients with an acute myocardial infarction. Clin Nutr. 2004 Aug;23(4):491-500.
6. Grundt H, Nilsen DW, Hetland Ø, Valente E, Fagertun HE. Activated factor 12 (FXIIa) predicts recurrent coronary events after an acute myocardial infarction. Am Heart J. 2004 Feb;147(2):260-6.
7. Aarsetøy H, Brügger-Andersen T, Hetland Ø, Grundt H, Nilsen DW. Long term influence of regular intake of high dose n-3 fatty acids on CD40-ligand, pregnancy-associated plasma protein A and matrix metalloproteinase-9 following acute myocardial infarction. Thromb Haemost. 2006 Feb;95(2):329-36.
8. Brügger-Andersen T, Aarsetøy H, Grundt H, Staines H, Nilsen DW. The long-term prognostic value of multiple biomarkers following a myocardial infarction.Thromb Res. 2008;123(1):60-6.
9. Aarsetøy H, Valente E, Reine A, Mansoor MA, Grundt H, Nilsen DW. Holotranscobalamin and methylmalonic acid as prognostic markers following an acute myocardial infarction. Eur J Clin Nutr. 2008 Mar;62(3):411-8. Epub 2007 Mar 7.

ELIGIBILITY:
Inclusion Criteria:

* Verified an acute myocardial infarction (MI) by World Health Organization criteria
* Age above 18 years
* Discontinuation of a regular supplementation of other fish-oil products
* Signed informed consent

Exclusion Criteria:

* Assumed noncompliance to protocol
* Expected survival < 2 y because of severe heart failure (New York Heart Association class IV), malignancy, or other reasons
* Ongoing gastrointestinal bleeding or verified stomach ulcer
* Thrombocytopenia or blood platelets < 100 x 10'9/L
* Liver insufficiency
* Participation in any other study
* Residence outside the recruitment area of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 1995-09; Primary Completion 1997-12 (Actual); Study Completion 2002-12 (Actual)

PRIMARY OUTCOMES:
Fatal and non-fatal cardiac events | 2 years
  Cardiac events were defined as cardiac death, resuscitation, recurrent myocardial infarction (MI) and unstable angina pectoris, presented as single or combined cardiac events. Revascularizations and death from other causes were also recorded.

SECONDARY OUTCOMES:
Serum lipids | One year
  Blood specimen were harvested at baseline [3-5 days post myocardial infarction (MI)] and repeated at 6 weeks, at 6 and 12 months follow-up. Serum cholesterol, high-density lipoprotein (HDL) - cholesterol and triacylglycerol were evaluated during follow-up.
Inflammation markers | One year
  Blood specimen were harvested at baseline [3-5 days post myocardial infarction (MI)] and repeated at 6 weeks, at 6 and 12 months follow-up. Several markers of inflammation [high-sensitivity C-Reactive Protein (CRP), CD40-Ligand] were evaluated during follow-up.
Coagulation markers | One year
  Blood specimen were harvested at baseline [3-5 days post myocardial infarction (MI)] and repeated at 6 weeks, at 6 and 12 months follow-up. Several markers of coagulation (fibrin monomer, fibrinogen, tissue factor, activated factor XII) were evaluated during follow-up.
Endothelial dysfunction | One year
  Blood specimen were harvested at baseline [3-5 days post myocardial infarction (MI)] and repeated at 6 weeks, at 6 and 12 months follow-up. Several markers of endothelial dysfunction (adhesion molecules, homocysteine) were evaluated during follow-up.
Oxidative stress | One year
  Blood specimen were harvested at baseline [3-5 days post myocardila infraction (MI)] and repeated at 6 weeks, at 6 and 12 months follow-up. Thiobarbituric acid Reactive Substances(TBARS), a marker of the oxidative burden of n-3 fatty acids, was evaluated during follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis WT Nilsen, PhD, Principal Investigator — Department of Medicine, the Division of Cardiology, the Central Hospital in Rogaland, Norway, and the University of Bergen, Norway
Locations (1):
- Central Hospital in Rogalanad, Stavanger, Norway

REFERENCES:
- [Background] Leaf A, Weber PC. Cardiovascular effects of n-3 fatty acids. N Engl J Med. 1988 Mar 3;318(9):549-57. doi: 10.1056/NEJM198803033180905. No abstract available. PMID 3277056
- [Background] Schmidt EB, Dyerberg J. Omega-3 fatty acids. Current status in cardiovascular medicine. Drugs. 1994 Mar;47(3):405-24. doi: 10.2165/00003495-199447030-00003. PMID 7514972
- [Background] Connor SL, Connor WE. Are fish oils beneficial in the prevention and treatment of coronary artery disease? Am J Clin Nutr. 1997 Oct;66(4 Suppl):1020S-1031S. doi: 10.1093/ajcn/66.4.1020S. PMID 9322583
- [Background] Sellmayer A, Witzgall H, Lorenz RL, Weber PC. Effects of dietary fish oil on ventricular premature complexes. Am J Cardiol. 1995 Nov 1;76(12):974-7. doi: 10.1016/s0002-9149(99)80276-8. PMID 7484845
- [Background] Bonaa KH, Bjerve KS, Straume B, Gram IT, Thelle D. Effect of eicosapentaenoic and docosahexaenoic acids on blood pressure in hypertension. A population-based intervention trial from the Tromso study. N Engl J Med. 1990 Mar 22;322(12):795-801. doi: 10.1056/NEJM199003223221202. PMID 2137901
- [Background] Harris WS. Fish oils and plasma lipid and lipoprotein metabolism in humans: a critical review. J Lipid Res. 1989 Jun;30(6):785-807. PMID 2677200
- [Background] Eritsland J, Arnesen H, Seljeflot I, Hostmark AT. Long-term metabolic effects of n-3 polyunsaturated fatty acids in patients with coronary artery disease. Am J Clin Nutr. 1995 Apr;61(4):831-6. doi: 10.1093/ajcn/61.4.831. PMID 7702027
- [Background] Jeppesen J, Hein HO, Suadicani P, Gyntelberg F. Triglyceride concentration and ischemic heart disease: an eight-year follow-up in the Copenhagen Male Study. Circulation. 1998 Mar 24;97(11):1029-36. doi: 10.1161/01.cir.97.11.1029. PMID 9531248
- [Derived] Naesgaard PA, Grundt H, Nordoy AF, Staines H, Nilsen DWT. Vitamin D Uptake in Patients Treated with a High-Dosed Purified Omega-3 Compound in a Randomized Clinical Trial Following an Acute Myocardial Infarction. Front Cardiovasc Med. 2017 Jul 24;4:41. doi: 10.3389/fcvm.2017.00041. eCollection 2017. PMID 28791297